CLINICAL TRIAL: NCT01155206
Title: Acute Regulation of Intestinal and Hepatic Lipoprotein Production by Glucagon
Acronym: Glucagon
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Gary Lewis, MD, University Health Network, Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 07-0394-A
Record Dates: First submitted 2008-06-25; First posted 2010-07-01 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2007-09

CONDITIONS: Diabetes
Keywords: glucagon,; high physiological dose and basal dose of glucagon; hepatic lipoprotein production,; free fatty acid; intestinal lipoprotein production; particle; glucagon affects production of fat in intestine and liver.
MeSH Terms: conditions — Diabetes Mellitus | interventions — Glucagon

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- high glucagon (Experimental): For one of the two studies to be performed in random order, the subject will receive an infusion of glucagon at a dose that has been shown to achieve high physiological plasma levels. The IV glucagon will be administered at a rate of 3ng/kg/min.
  Interventions: Drug: glucagon
- low glucagon (Experimental): For one of the two studies to be performed in random order, the subject will receive an infusion of glucagon at a low rate that is designed to mimic basal plasma glucagon concentration. The IV glucagon will be administered at a rate of 0.65ng/kg/min.
  Interventions: Drug: glucagon

INTERVENTIONS:
Drug: glucagon — glucagon 3ng/kg/min
  Other Names: glucagon 0.65ng/kg/min

SUMMARY:
Insulin resistant states are characterized by hepatic lipoprotein (VLDL) particle overproduction. Numerous hormonal and nutritional factors are known to influence hepatic lipoprotein particle production, including insulin and free fatty acids (FFA). In contrast to the liver, the intestine has traditionally been viewed as a 'passive' organ with respect to lipoprotein production, with intestinal lipoprotein particle production determined mainly by the amount of fat ingested and absorbed. Glucagon plays a key role in the regulation of carbohydrate and fatty acid metabolism and has recently been shown for the first time to regulate hepatic lipoprotein production in mice. Ours will be the first study to investigate the effect of glucagon on hepatic and intestinal lipoprotein production in humans.

DETAILED DESCRIPTION:
Potential role of glucagon in intestinal and hepatic lipoprotein production. Although glucagon, the main hormone that opposes insulin action, is known to exert profound effects on carbohydrate (stimulation of hepatic glucose production) and fatty acid metabolism (stimulation of hepatic b-oxidation and ketogenesis), its potential role in the regulation of lipoprotein metabolism has been largely overlooked and the mechanism whereby glucagon modulates hepatic lipid metabolism in humans has not previously been examined. Longuet et al recently showed that glucagon receptor (Gcgr) signaling is essential for control of hepatic lipid homeostasis in mice (44). They showed that Gcgr-/- mice exhibit higher plasma TG levels and increased hepatic TG production compared to littermate controls. Conversely, glucagon administration to wildtype mice decreased hepatic lipid production and plasma TGs. A combination of microarray and RealTime PCR analyses demonstrated that a period of fasting increased the expression of genes regulating fatty acid b-oxidation in +/+ but not in Gcgr-/- mice. Furthermore, exogenous glucagon administration mimicked the increase in expression of enzymes involved in b-oxidation during fasting in +/+ mice. Enzymes involved in fatty acid synthesis were not regulated by exogenous glucagon. Gcgr-/- mice were much more susceptible to the accumulation of lipids in the liver, known to be associated with the development of non-alcoholic steatohepatitis. To date, glucagon regulation of intestinal lipoprotein production has not been examined in animals or humans.

There is convincing evidence from mouse studies that glucagon plays a major role in the regulation of hepatic lipoprotein production and may also play a role in intestinal lipoprotein assembly and secretion. Ours will be the first study to examine the role of glucagon in hepatic and intestinal lipoprotein production in humans. Since inhibition of glucagon receptor activity is currently being explored as a therapeutic approach for the treatment of Type 2 diabetes, our study will provide important information regarding potential implications of this therapeutic approach for control of lipid homeostasis and general metabolic health.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged 18 to 40 years
2. Body mass index 20 kg/m2 to 25 kg/m2
3. Hemoglobin above 130g/L.
4. Normal glucose tolerance in response to a 75g, 2-hr OGTT

Exclusion Criteria:

1. Subject has a history of hepatitis/hepatic disease that has been active within the previous two years.
2. Any significant active (over the past 12 months) disease of the gastrointestinal, pulmonary, neurological, renal (Cr > 1.5 mg/dL), genitourinary, hematological systems, or has severe uncontrolled treated or untreated hypertension (sitting diastolic BP > 100 or systolic > 180) or proliferative retinopathy
3. Fasting blood glucose > 6.0 mmol/l or known diabetes.
4. Any history of a MI or clinically significant, active, cardiovascular history including a history of arrhythmia's or conduction delays on ECG, unstable angina, or decompensated heart failure.
5. Any laboratory values: AST > 2x ULN; ALT > 2x ULN TSH > 6 mU/l
6. Current addiction to alcohol or substances of abuse as determined by the investigator.
7. Mental incapacity, unwillingness or language barrier precluding adequate understanding or cooperation
8. Taking any prescription or non-prescription medications at the time of the study
9. Having donated blood three months prior to and three months post study procedures
10. A pregnancy test will be performed 1 to 3 days prior to each study in all female subjects. Those who test positive for pregnancy will be excluded.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2009-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Triglyceride-rich lipoprotein production rate | 0-10 hours

CONTACTS AND LOCATIONS:
Overall Officials: Gary F Lewis, MD, Principal Investigator — University Health Network, Toronto General Hospital
Locations (1):
- University Health Network, Toronto General Hospital, Toronto, Ontario, Canada